CLINICAL TRIAL: NCT02495675
Title: Effects of Treatment With High Flow Nasal Cannulas on Respiratory Pattern and Work of Breathing Among Healthy Subjects
Acronym: HDWOBSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IUCPQ-HDWOBSS
Record Dates: First submitted 2015-06-04; First posted 2015-07-13 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- No flow (No Intervention): Subjects will be spontaneously breathing in room air with no flow.
- Conventional flow via nasal prongs (Experimental): Subjects will be breathing with nasal prongs delivering 5 L/min of air (inspired fraction of oxygen: 0.21)
  Interventions: Device: Conventional flow via nasal prongs
- High flow nasal cannulas 20 L/min (Experimental): Subjects will be breathing with high flow nasal cannulas delivering 20 L/min with an inspired fraction of oxygen of 0.21.
  Interventions: Device: High flow nasal cannulas
- High flow nasal cannulas 40 L/min (Experimental): Subjects will be breathing with high flow nasal cannulas delivering 40 L/min with an inspired fraction of oxygen of 0.21.
  Interventions: Device: High flow nasal cannulas
- High flow nasal cannulas 60 L/min (Experimental): Subjects will be breathing with high flow nasal cannulas delivering 60 L/min with an inspired fraction of oxygen of 0.21.
  Interventions: Device: High flow nasal cannulas

INTERVENTIONS:
Device: High flow nasal cannulas — Comparison of different flow levels
  Other Names: Airvo 2; Ficher and Paykel HealthCare
  Arms: High flow nasal cannulas 20 L/min; High flow nasal cannulas 40 L/min; High flow nasal cannulas 60 L/min
Device: Conventional flow via nasal prongs — Low flow of air delivered through conventional nasal prongs
  Arms: Conventional flow via nasal prongs

SUMMARY:
This study evaluates the work of breathing among healthy subjects under various conditions of treatment with high flow nasal cannulas. Ten subjects will be included. The design of this study is a cross over of five treatment periods with different flow settings.

DETAILED DESCRIPTION:
High flow oxygen therapy (HFOT) is a promising technique increasingly used in the management of acute respiratory failure. In hospitalised hypoxemic patients, recent clinical evidence showed that HFOT can reduce endotracheal intubation and reduce mortality. Physiologically, the HFOT causes a decrease in respiratory rate and minute-ventilation and may be associated with a decrease in carbone dioxyde arterial pressure. It is possible that these effects are associated with decreased work of breathing, which could explain some of the benefits in terms of comfort and efficiency.

The objective of this research is to evaluate the impact of a wash-out of anatomical dead space by high flow nasal cannulas on respiratory parameters and on the work of breathing among healthy subjects. The investigators will evaluate the baseline status in room air, and then compare it with four different levels of flow. The primary endpoint will be the work of breathing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Written and informed consent

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Subject enrolled in another study excluding co-enrolment;
* Cardio-vascular or respiratory disease;
* History of ear nose and throat disease (i.e. surgery, epistaxis, trauma), eso-gastric disease (i.e. esophageal varices, digestive haemorrhage), rheumatologic or neurologic disease possibly interfering with the design of the study;
* Subject feeling nauseous or under recent fed condition (<1h).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Work of breathing | 10 minutes
  Work of breathing at the end of each period is calculated from the measurement of esophageal pressure and tidal volume (composite outcome).

SECONDARY OUTCOMES:
Esophageal pressure-time product | 10 minutes
  Measured at the end of each period
Tidal Volume | 10 minutes
  Measured at the end of each period
Comfort of breathing | 10 minutes
  Subjective evaluation at the end of each period
Blood gases | 10 minutes
  Arterial or capillary blood gases at the end of each period
Dyspnea | 10 minutes
  Evaluation on a borg scale at the end of each period
Respiratory Rate | 10 minutes
  Measured at the end of each period
End-tidal carbon dioxide | 10 minutes
  Measured at the end of each period
Heart rate | 10 minutes
  Measured at the end of each period
Oxygen saturation | 10 minutes
  Measured at the end of each period

CONTACTS AND LOCATIONS:
Overall Officials: François Lellouche, MD, PhD, Study Director — Fondation IUCPQ
Locations (1):
- Centre de Recherche de l'IUCPQ, Québec, Quebec, Canada

REFERENCES:
- [Derived] Delorme M, Bouchard PA, Simon M, Simard S, Lellouche F. Physiologic Effects of High-Flow Nasal Cannula in Healthy Subjects. Respir Care. 2020 Sep;65(9):1346-1354. doi: 10.4187/respcare.07306. Epub 2020 Apr 14. PMID 32291309